CLINICAL TRIAL: NCT07299734
Title: Assessing the Feasibility and Safety of a Combined Closed Loop Functional Electrical Stimulation and Augmented Reality System for Individuals With Cervical Spinal Cord Injury
Brief Title: Feasibility and Safety of a Combined Augmented Reality and Functional Electrical Stimulation System
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Training Platform for Trials Leveraging Existing Networks (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 25-5898
Record Dates: First submitted 2025-11-25; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-11

CONDITIONS: Cervical Spinal Cord Injury
Keywords: Cervical spinal cord injury; Augmented reality; Functional electrical stimulation; Neuromodulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single group (Experimental): Participants will go through 1 screening session, 20 experimental sessions (2 sessions per week for 10 weeks), 1 discharge assessment, and 1 follow up assessment (one month after the last experimental session).
  Interventions: Device: AR + FES

INTERVENTIONS:
Device: AR + FES — Within each one-hour experimental session, participants will interact with different objects (e.g. block, credit card, marble). They will be wearing an augmented reality (AR) headset and electrodes will be placed over finger flexors, thumb flexors and finger extensors muscles. The AR headset will track hand posture and use the difference between the actual posture and a target posture to regulate functional electrical stimulation (FES) delivered via the electrodes.

SUMMARY:
Cervical spinal cord injury (cSCI) can result in substantial loss of upper-limb function, with associated socio-economic impact on affected individuals and the healthcare system. Evidence suggests that non-invasive neuromodulation such as functional electrical stimulation (FES) therapy can contribute to regaining upper-limb function, which is a top priority for this population. This pilot study will involve individuals with cSCI using a device that combines augmented reality (AR) and functional electrical stimulation (FES) for 20, one-hour sessions over a 10-week period. The sessions will include upper-limb rehabilitation where individuals will interact with different objects with the aid of the AR +FES system. The primary objective is to assess safety and feasibility, measured by the absence of serious adverse events and participants' ability to independently set up and use the system. Secondary objectives include adherence to the intervention and user feedback through structured interviews. Exploratory outcomes will examine preliminary efficacy using clinical measures such as the Spinal Cord Independence Measure (SCIM) and the Graded Redefined Assessment of Strength, Sensation and Prehension (GRASSP).

ELIGIBILITY:
Inclusion Criteria:

* Chronic cervical SCI
* Any level or severity of cervical SCI, traumatic or non-traumatic
* Can carry out object manipulations but with visible impairment (i.e., 5-25 on the GRASSP Prehension Performance sub-score).

Exclusion Criteria:

* Any disease or injury other than the SCI that may be affecting grasping performance.
* Individuals with any self-reported FES contraindications (pacemakers, implantable defibrillator, implanted neurostimulation device, metallic implants in the stimulated areas, cardiac conditions, epilepsy, uncontrolled seizures, wounds or fractures on the target limb)
* Inability to understand the study procedures
* Muscles do not respond to FES to produce grasping movements
* Currently participating in another upper limb rehabilitation intervention study (regular physical and occupational therapy is permitted).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Week 1 to week 14.
  Presence of adverse and serious adverse events. These will be recorded during each session. The criterion for success is no study-related serious adverse events and no study-related adverse events that cannot be alleviated by stopping electrical stimulation.
Feasibility - Set-up time | During experimental sessions from week 1 to week 10.
  The study will track independence with the system by assessing set-up time.
Feasibility - Assistance required. | During experimental sessions from week 1 to week 10.
  The study will track independence with the system by assessing the number of times assistance is requested.

SECONDARY OUTCOMES:
Adherence | During experimental sessions from week 1 to week 10.
  Number of missed sessions.
User feedback | Discharge assessment at week 10.
  Structured and semi-structured interviews.

OTHER OUTCOMES:
Graded Redefined Assessment of Strength, Sensation and Prehension | Baseline (week 0), discharge (week 10) and follow-up (week 14) assessments.
  Hand function assessment.
Spinal Cord Independence Measure | Baseline (week 0), discharge (week 10) and follow-up (week 14) assessments.
  Questionnaire about independence on daily tasks.

CONTACTS AND LOCATIONS:
Overall Officials: José Zariffa, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Lyndhurst Centre, Toronto Rehabilitation Institute - University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified coded study data may be used or shared with other researchers for future studies. Directly identifying information will be replaced by a number, which will be applied to the study data. The participant key matching the code to the participant will be kept by the UHN study team. This may include storing the coded study data in controlled-access databases or open access, publicly accessible databases.